CLINICAL TRIAL: NCT05060146
Title: Prevention of Pneumococcal Infections: Impact Collaborative Medico-pharmaceutical Care Structured to Improve Vaccination Coverage of Patients at Risk.
Acronym: OPTIVACC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: PHRC-I/2019/FD-01; 2020-A01581-38 (Other: ANSM)
Record Dates: First submitted 2021-09-07; First posted 2021-09-29 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-10

CONDITIONS: Streptococcus Pneumoniae Infection
MeSH Terms: conditions — Pneumococcal Infections

STUDY DESIGN:
Intervention Model Description: Step wedge
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention)
- Structured medico-pharmaceutical collaboration (Experimental)
  Interventions: Other: Structured medico-pharmaceutical collaboration

INTERVENTIONS:
Other: Structured medico-pharmaceutical collaboration — Reconciliation of drug treatments; Writing of the prescription for discharge from hospital for the pneumococcal vaccine; Pharmaceutical interview at discharge; Drafting of the discharge letter and transmission to the attending physician; Writing of the pharmaceutical discharge letter and transmission to the pharmacist; Pharmaceutical dispensing in the pharmacy; Administration of the vaccine by the attending physician or a nurse at home.
  Arms: Structured medico-pharmaceutical collaboration

SUMMARY:
In France, Streptococcus pneumoniae is the leading agent bacterial involved in community lung disease and meningitis. The frequency of these infections and their mortality increase significantly in those at risk such as patients with certain chronic diseases, immunocompromised or on immunosuppressive therapy. This population, despite regular monitoring, has a limited pneumococcal vaccine coverage of around 20%. By carrying out a reconciliation of treatments upon admission to hospital, the clinical pharmacist can detect those without up to date pneumococcal vaccination status. The goal of this management is to make the patient aware of the need for vaccination and organization upon return home. Thus, this limited pneumococcal vaccination coverage would benefit from intervention by regional clinical pharmacy activities. The study investigators want to study the impact of a structured medico-pharmaceutical collaboration on pneumococcal vaccination of patients with risk on discharge from hospital. The investigators hypothesize that this collaboration in patients at risk of infection with pneumococcus could significantly increase their anti-pneumococcal vaccination coverage

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed oral consent
* The patient must be a member or beneficiary of a health insurance plan
* The patient is admitted to full hospitalization in a surgical or medical department.
* The patient will benefit from a reconciliation of drug treatments.
* The patient is considered at risk of pneumococcal infection according to the recommendations of March 2017 of the High Council of Public Health (HCSP)
* Pneumococcal vaccination is not up to date according to the HCSP 2017 recommendations.

Exclusion Criteria:

* The subject is participating in a category 1 interventional study
* The patient has participated in a category 1 trial within the previous 3 months or is in a period of exclusion determined by a previous study
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is not in a fit state to express consent
* The patient is pregnant, parturient or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2024-06-12 (Actual); Study Completion 2024-06-12 (Actual)

PRIMARY OUTCOMES:
Full vaccination coverage (2 doses) between groups | 6 months after discharge
  Yes/No, confirmed by the administrator

SECONDARY OUTCOMES:
Full vaccination coverage (2 doses) between groups, stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | 6 months after discharge
  Yes/No, confirmed by the administrator
Partial vaccination coverage (1st dose only) between groups and stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | 6 months after discharge
  Yes/No, confirmed by the administrator
Record of both vaccines being dispensed by the pharmacy between groups and stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | 6 months after last follow-up visit
  Yes/No according to Système national d'information inter-régimes de l'Assurance maladie (SNIIRAM) database
Concordance between vaccines dispensed and vaccines recorded in the SNIRRAM database between groups and stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | 6 months after discharge
  Yes/No
Prescription of vaccines at discharge by the doctor between groups and stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | at discharge (average 5 days after hospitlization)
  Yes/No
Notification of requirement for vaccine between groups and stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | at discharge (average 5 days after hospitlization)
  Yes/No
Transmission of letter highlighting the absence of vaccination by the pharmacy to the patient's doctor between groups and stratified by type of establishment (University hospital vs hospital) and by service (Medicine vs Surgery) | at discharge (average 5 days after hospitlization)
  Yes/No

CONTACTS AND LOCATIONS:
Overall Officials: Florent Dubois, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (9):
- France (9):
  - CH Alès Cévennes, Alès
  - CH de Bagnols sur Cèze, Bagnols-sur-Cèze
  - CH de Montauban, Montauban
  - CHU de Montpellier, Montpellier
  - CHU de Nimes, Nîmes
  - CH de Perpignan, Perpignan
  - CH Comminges Pyrénées, Saint-Gaudens
  - CH du Bassin de Thau, Sète
  - CHU de Toulouse, Toulouse

REFERENCES:
- [Result] Dubois F, Champiot-Bayard E, Cireasa B, Loubet P, Vallat J, Bonnet J, Jacob V, Puyo P, Pinzar I, Theret S, Dubois E, Peus E, Giraudon L, Roux-Marson C, Fabbro-Peray P, Leguelinel-Blache G, Kinowski JM. Prevention of pneumococcal infections: Impact of structured medico-pharmaceutical collaborative management to improve vaccination coverage of at-risk patients (OPTIVACC study): Protocol for a multicenter randomized stepped -wedge study. Contemp Clin Trials Commun. 2025 Feb 15;44:101462. doi: 10.1016/j.conctc.2025.101462. eCollection 2025 Apr. PMID 40065836